CLINICAL TRIAL: NCT02278302
Title: Placebo-controlled, Randomized, Double-blind Study Comparing the Effect of a Combination of 200 mg Dipyridamole With Sustained Release and 25 mg Acetyl Salicylic Acid (Aggrenox®) on the Performance Relevant to Safety and on the General Condition of Volunteers and 10 Days of Treatment Alone and in Combination With Alcohol (Study no. 591002)
Brief Title: Study to Compare the Effect of a Combination of Dipyridamole With Sustained Release and Acetyl Salicylic Acid (Aggrenox®) on the Performance Relevant to Safety and on the General Condition of Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9.135
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Aspirin, Dipyridamole Drug Combination; Ethanol

ARMS (2):
- Aggrenox® (Experimental): treatment alone or in combination with Ethanol
  Interventions: Drug: Aggrenox®; Other: Ethanol
- Placebo (Placebo Comparator): treatment alone or in combination with Ethanol
  Interventions: Drug: Placebo; Other: Ethanol

INTERVENTIONS:
Drug: Aggrenox®
  Arms: Aggrenox®
Drug: Placebo
  Arms: Placebo
Other: Ethanol

SUMMARY:
Study to investigate whether psychomotor performance which is necessary for safety driving a car or operating machinery and safely participating in daily life is changed by Aggrenox®. Also to investigate whether Aggrenox® impairs performance in combination with alcohol more than alcohol alone. Derived from this: Statement on whether a warning for drivers is necessary

ELIGIBILITY:
Inclusion Criteria:

* Race: Caucasian
* Men and women aged between 40 and 65 years
* Written and spoken command of German
* Ability to understand the nature and significance of the study
* Written informed consent to participate in the study

Exclusion Criteria:

* Acute disease at the beginning of the study
* Any chronic disease in particular:

  * Diseases for which the administration of the test drug was contraindicated:
  * Severe coronary heart disease (e.g. unstable angina pectoris or recent myocardial infarction)
  * Subvalvular aortic stenosis or hemodynamic instability, myocardial decompensation
  * Severe hypotension, hypotonic collapse
  * Any other cardiac disease (or case history of)
  * Chronic obstructive lung disease
  * Hepatic and renal dysfunction
  * Diseases of the gastrointestinal tract
  * Mental or neurologic diseases
  * Alcoholism, alcohol abuse
  * Case history of clinically relevant allergies (particularly against one of the ingredients of the test substance incl. paracetamol)
  * Participation in another clinical study during the last two months preceding the study
* Women while pregnant or breastfeeding
* Women of childbearing age without safe contraception
* Psychotropic drugs during the last four weeks before the beginning of and during the study
* taking other medicaments regularly during the last two weeks before the beginning of and during the study (except for oral contraceptives, hormone replacement in women)
* Body weight outside the Body-Mass-Index (BMI) +- 4
* Habits of life style having a presumable negative effect on the results of the performance test (e.g. shift work, extreme sports, blood donation within the last 4 weeks, > 8 cups/glasses of caffeine-containing beverages/day, > 40 g alcohol/day, >40 cigarettes/day)
* positive or no drug screening for barbiturates, benzodiazepines, tricyclic antidepressants and cannabinoids, amphetamines, cocaine, opiates
* Persons having been detained in an institution by judicial or official order
* Persons incapacitated or placed under provisional guardianship

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 1999-08; Primary Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
Change in safety relevant performance in the steady state represented and scored by five psychomotor tests | up to day 11
  motor coordination, reaction under stress, concentration, vigilance, precision and visual orientation

SECONDARY OUTCOMES:
Change in general condition rated on 4-point scales | up to day 11
Change in motor coordination by means of psychomotor test (2HAND) | up to day 11
Change in reaction under stress by means of psychomotor test (DT) | up to day 11
Change in vigilance by means of psychomotor test (VIGIL) | up to day 11
Change in concentration by means of psychomotor test (SIGNAL) | up to day 11
Change in precision and visual orientation by means of psychomotor test (TAVT33) | up to day 11
Number of subjects with adverse events | up to 25 days
Number of subjects with abnormal changes in laboratory parameters | up to day 11
Number of subjects with abnormal changes in vital parameters | up to day 11
  Blood Pressure, Pulse Rate, Body temperature